CLINICAL TRIAL: NCT06727617
Title: Serplulimab Plus Chemoradiotherapy vs Chemoradiotherapy as Adjuvant Treatment for Postoperative Cervical Cancer Patients With Multiple Risk Factors: A Randomized, Open-Label, Phase II Clinical Trial
Brief Title: Serplulimab With Chemoradiotherapy for Postoperative Cervical Cancer With Risk Factors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20241188A
Record Dates: First submitted 2024-12-01; First posted 2024-12-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancers
Keywords: cervical cancer; high risk; immunotherapy; radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serplulimab plus chemoradiotherapy group (Experimental): Serplulimab plus chemoradiotherapy group
  Interventions: Drug: Serplulimab; Drug: Chemotherapy; Radiation: radiotherapy
- chemoradiotherapy group (Placebo Comparator): chemoradiotherapy group
  Interventions: Drug: Chemotherapy; Radiation: radiotherapy

INTERVENTIONS:
Drug: Serplulimab — intravenous infusion of 300 mg, administered every 3 weeks as one cycle, on the first day of each cycle, with a maximum treatment duration of 2 years (up to 35 treatment cycles)
  Arms: Serplulimab plus chemoradiotherapy group
Drug: Chemotherapy — Cisplatin: Administered by intravenous infusion during concurrent chemoradiotherapy at a dose of 30-40 mg/m² once weekly for only 5-6 treatment cycles; during sequential chemoradiotherapy, administered at 60-75 mg/m² on the first and second days of each cycle, once every 3 weeks (21 days) for only 4 treatment cycles.
  Paclitaxel: Nab-paclitaxel administered by intravenous infusion at a dose of 135-175 mg/m² on the first day of each cycle, once every 3 weeks (21 days) for only 4 treatment cycles.
Radiation: radiotherapy — Pelvic external beam radiation therapy at a dose of 1.8 Gy per fraction or 2 Gy per day, 5 times per week, with a total dose of 45-50 Gy.

SUMMARY:
A Phase II Study of Serplulimab Plus Chemoradiotherapy as Adjuvant Treatment for Postoperative Cervical Cancer with Multiple Risk Factors

DETAILED DESCRIPTION:
This study is a randomized, controlled, open-label, Phase II clinical trial designed to enroll patients with at least two risk factors (risk factors: lymph node metastasis, positive parametrial or resection margins, lymphovascular space invasion, or deep stromal invasion) following radical surgery for cervical cancer. The study aims to evaluate the efficacy and safety of Serplulimab in combination with chemoradiotherapy compared to chemoradiotherapy alone as adjuvant treatment. Patients must be deemed suitable for cisplatin or carboplatin plus nab-paclitaxel treatment as determined by the investigator. The choice between carboplatin and cisplatin will be based on the clinical judgment of the investigator. Eligible patients will be randomized in a 1:1 ratio to one of the following treatment arms: patients receiving Serplulimab plus chemoradiotherapy as adjuvant treatment (experimental group) or patients receiving chemoradiotherapy alone as adjuvant treatment (control group). The study is expected to enroll 67 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the clinical study: Fully understand and be informed about the study, and sign the informed consent form (ICF); willing to comply with and capable of completing all trial procedures.
* Female aged ≥18 years and ≤65 years at the time of signing the ICF.
* ECOG PS score of 0 or 1.
* Positive PD-L1 status (CPS ≥1).
* Diagnosed with cervical squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma.
* FIGO (International Federation of Gynecology and Obstetrics) stage of IB1, IB2, IIA1, or IIA2, and patients judged by the investigator to benefit from radical surgery and/or adjuvant therapy.
* Have undergone radical hysterectomy (Piver classification) and pelvic lymphadenectomy of type II or III.
* Postoperative pathological examination confirms at least two adverse factors, which may include: Lymph node metastasis; Positive parametrial or positive resection margins; Lymphovascular space invasion; Deep stromal invasion;
* Patients must meet the following hematological, renal, and liver function criteria: Absolute neutrophil count of at least 1.5 × 10⁹/L; Platelet count of at least 100 × 10⁹/L; Total bilirubin, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) levels not exceeding 1.5 times the upper limit of normal; Creatinine levels not exceeding the upper limit of normal.
* Female participants must have a negative serum pregnancy test within 14 days prior to treatment and agree to use effective contraception during the treatment period and for 6 months afterward; breastfeeding is prohibited during treatment.
* Willing and able to comply with the trial and follow-up procedures.

Exclusion Criteria:

* Patients with unresectable residual tumors.
* Histologically confirmed diagnosis of cervical small cell carcinoma (neuroendocrine) or mucinous adenocarcinoma.
* Patients who have previously received pelvic radiotherapy.
* History of other untreated malignant tumors within the past 5 years, except for cured basal cell carcinoma of the skin or carcinoma in situ.
* Presence of any active or known autoimmune disease.
* History of inflammatory/autoimmune diseases requiring steroid treatment, or currently suffering from inflammatory/autoimmune diseases that require steroid treatment.
* Diseases requiring systemic treatment with corticosteroids or other immunosuppressive agents within 14 days prior to randomization.
* History of thromboembolic events (venous or arterial) occurring within 6 months prior to enrollment.
* Poorly controlled clinical symptoms or conditions related to heart disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
DFS | through study completion, an average of 1 year
  The time from the date of random assignment to the first occurrence of locoregional failure, DM, second primary tumor, or death from any cause.

SECONDARY OUTCOMES:
OS | through study completion, an average of 1 year
  The time from random assignment to death because of any cause.
RFS | through study completion, an average of 1 year
  The time from random assignment to death because of any recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Maobin Meng, Dr., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China